CLINICAL TRIAL: NCT02735070
Title: Phase III Study Comparing Coristina® D to Resfenol® in the Symptomatic Treatment of Common Cold
Brief Title: Study Comparing Coristina® D to Resfenol® in the Symptomatic Treatment of Common Cold
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brainfarma Industria Química e Farmacêutica S/A (Industry)
Collaborators: Techtrials Pesquisa e Tecnologia Ltda (Unknown); Pharmagenix (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Coristina® d
Record Dates: First submitted 2016-03-18; First posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Cold
Keywords: Common cold treatment
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corisitina D (Experimental): The patient will use the medication 4 times a day - orally The tablets of Coristina® d contain 400 mg acetylsalicylic acid, dexchlorpheniramine 1 mg, 10 mg phenylephrine, and 30 mg of caffeine. Coristina® d is indicated as an analgesic, antipyretic, antiallergic, and nasal congestion for the treatment of the symptoms of influenza and common cold.
  Interventions: Drug: Coristina d
- Resfenol (Active Comparator): The patient will use the medication 4x / day - orally Resfenol® drug acts against the symptoms of colds and flu, such as nasal congestion, runny nose, fever, headache, muscle pain and other symptoms. The capsules containing 400mg of paracetamol, 4 mg chlorpheniramine and 4mg phenylephrine.
  Interventions: Drug: Resfenol

INTERVENTIONS:
Drug: Resfenol — Patients should take the study medication without breaking or chewing together with a cup containing approximately 200 ml of water. The patient should ingest the study drug after fasting for at least 30 minutes.
  Arms: Resfenol
Drug: Coristina d — Patients included in the study will take the drugs 4 times a day, orally. Patients should take the study medication without breaking or chewing together with a cup containing approximately 200 ml of water. The patient should ingest the study drug after fasting for at least 30 minutes.
  Arms: Corisitina D

SUMMARY:
The primary objective of this study is to evaluate the non-inferiority of Coristina® d in the symptomatic treatment of the common cold compared to Resfenol® comparator.

DETAILED DESCRIPTION:
Eligible patients must sign the informed consent form and they will be between 18 and 60 years old and common cold symptoms for no more than 72 hours.

It will be recruited for this study 366 patients, 183 patients per group. It is estimated that the total number of patients can be recruited in 4 to 6 months from the regulatory approval of the study.

The patient will stay in the study approximately 7 to 10 days (including screening visit / randomization, telephone contact in 3 to 5 days after randomization and final visit from 1 to 3 days after last dose).

Study medication (Coristina d and Resfenol) will be provided by the sponsor and will be appropriately labeled for the clinical study, containing the sponsor information, the trial identification, expiration date, batch and storage conditions

ELIGIBILITY:
Inclusion Criteria:

1. Sign and date the informed consent form;
2. Age between 18 and 60 years old;
3. Symptoms of common cold not exceeding 72 hours must be present;
4. It will be considered symptoms of the common cold the presence of at least 2 of the 10 symptoms following: runny nose, sneezing, nasal congestion, headache, myalgia, throat discomfort or sore throat, hoarseness, cough or fever. Each of the symptoms listed above will receive a score by Likert scale (no symptom = 0, mild symptoms = 1, moderate symptoms = 2, intense symptoms = 3). The minimum total is 0 and maximum one is 30, which included patients with score higher or equal to 4 points.

Exclusion Criteria:

1. Presence of suggestive symptoms or prior diagnosis requiring regular and continuous treatment of allergic rhinitis or asthma in the last 2 years;
2. Chronic disease of any kind that is contraindicate the participation of the patient based on the opinion of investigator;
3. Hypersensitivity or contraindication to use of components of the study medications;
4. Pregnant or women of childbearing age without adequate contraception;
5. Use of other anti-influenza drugs programmed during the study or for the last 5 days;
6. Regular active smokers (more than 3 cigarettes a day);
7. Participation in another clinical study in less than one year (unless justified benefit by the investigator).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 366 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Global Evaluation from 1 to 3 days after last dose | From 1 to 3 days after the last dose
  The primary outcome will be the global evaluation from investigator to be done from 1 to 3 days after the last dose.

SECONDARY OUTCOMES:
Likert Scale for symptons | From the screening until 1 to 3 days after the last dose
  It will be used a Likert Scale to evaluate the intensity of cold symptoms. It will be used at screening, between 3-5 days of randomization and between 1 to 3 days after the last dose.
Sleep Questionnaire | From the screening until 1 to 3 days after the last dose
  It will be used a Sleep questionnaire to evaluate the sleep quality. It will be used at screening, between 3-5 days of randomization and between 1 to 3 days after the last dose.
Daily Activities | From the screening until 1 to 3 days after the last dose
  It will be used a daily activities questionnaire to evaluate the physical and mental disposition on the routine daily activities. It will be used at screening, between 3-5 days of randomization and between 1 to 3 days after the last dose.
Adverse Events | From the randomization until 1 to 3 days after the last dose
  It will be evaluated and monitored the adverse events in order to assess the patient safety. It will be evaluated from randomization up to 1-3 days after last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Márcio Antônio Pereira, Dr., Principal Investigator — MAP Clínica de Endocrinologia Ltda; Amanda Faulhaber, Dr., Principal Investigator — Pesquisare Saude S/S Ltda; Clóvis Eduardo S Galvão, Dr., Principal Investigator — Instituto de Pesquisa Clínica e Medicina Avançada - IMA; Antônio Carlos da Silva, Dr., Principal Investigator — Clinilive; Paula YU Tokunaga, Dr., Principal Investigator — Centro de Estudos Clínicos do Interior Paulista - CECIP; Carlos I Filho, Dr., Principal Investigator — Unidade de Pesquisa Clínica do Centro de Medicina Reprodutiva Dr.Carlos Isaia Filho Ltda.; Durval C Kraychete, Dr., Principal Investigator — CTD Dor Clinica de Diagnostico e Terapia da Dor Ltda; Lívia FA Oliveira, Dr., Principal Investigator — Universidade Federal do Triângulo Mineiro - Núcleo de Estudos Clínicos; Flávio Sano, Dr., Principal Investigator — Departamento Centro de Estudos do Hospital Nipo-Brasileiro; Martti A Antila, Dr., Principal Investigator — Clínica de Alergia Martti Antila S/C Ltda

IPD SHARING:
Plan to Share IPD: Yes
The data that will be collected are: demographics data; medical history, disease characteristics; Likert scale; physician and patient perception about the study treatment; Sleep Questionnaire; evaluation for daily activities willingness; Safety Assessments; Vital Signs and Physical Examination; additional tests; Adverse Events.
  All data collected for the study will be recorded, stored and retrieved through electronic case report form designed specifically for this study.
  All information will be inserted in a database. All data collected for the study will be analyzed centrally by independent scientific consulting company designated for this purpose. The publication of the overall results of the study will be coordinated by the sponsor. The responsibility for the content of the publications will be shared between the sponsor and co-authors, who will participate in the review of the content and give consent for publication.

REFERENCES:
- [Result] De Sutter AI, van Driel ML, Kumar AA, Lesslar O, Skrt A. Oral antihistamine-decongestant-analgesic combinations for the common cold. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD004976. doi: 10.1002/14651858.CD004976.pub3. PMID 22336807
- [Result] Allan GM, Arroll B. Prevention and treatment of the common cold: making sense of the evidence. CMAJ. 2014 Feb 18;186(3):190-9. doi: 10.1503/cmaj.121442. Epub 2014 Jan 27. No abstract available. PMID 24468694
- [Result] Picon PD, Costa MB, da Veiga Picon R, Fendt LC, Suksteris ML, Saccilotto IC, Dornelles AD, Schmidt LF. Symptomatic treatment of the common cold with a fixed-dose combination of paracetamol, chlorphenamine and phenylephrine: a randomized, placebo-controlled trial. BMC Infect Dis. 2013 Nov 22;13:556. doi: 10.1186/1471-2334-13-556. PMID 24261438
- [Result] Mizoguchi H, Wilson A, Jerdack GR, Hull JD, Goodale M, Grender JM, Tyler BA. Efficacy of a single evening dose of syrup containing paracetamol, dextromethorphan hydrobromide, doxylamine succinate and ephedrine sulfate in subjects with multiple common cold symptoms. Int J Clin Pharmacol Ther. 2007 Apr;45(4):230-6. doi: 10.5414/cpp45230. PMID 17474541
- [Result] Common Cold Collaborative Group; Robert M, Llorens M, Garcia E, Luria X. Efficacy and tolerability of ebastine 10 mg plus pseudoephedrine 120 mg in the symptomatic relief of the common cold. Eur J Intern Med. 2004 Jul;15(4):242-247. doi: 10.1016/j.ejim.2004.03.009. PMID 15288679
- [Result] Bula Coristina d (Nov 2012, atualizada em 2014).
- [Result] Micromedex novembro de 2015: ácido acetilsalicílico Micromedex novembro de 2015: dexclorfeniramina
- [Result] Bantz EW, Dolen WK, Chadwick EW, Nelson HS. Chronic chlorpheniramine therapy: subsensitivity, drug metabolism, and compliance. Ann Allergy. 1987 Nov;59(5):341-6. PMID 3688558
- [Result] Munch EP, Soborg M, Norreslet TT, Mygind N. A comparative study of dexchlorpheniramine maleate sustained release tablets and budesonide nasal spray in seasonal allergic rhinitis. Allergy. 1983 Oct;38(7):517-24. doi: 10.1111/j.1398-9995.1983.tb02361.x. PMID 6139040
- [Result] Pastorello EA, Ortolani C, Gerosa S, Pravettoni V, Codecasa LR, Fugazza A, Zanussi C. Antihistaminic treatment of allergic rhinitis: a double-blind study with terfenadine versus dexchlorpheniramine. Pharmatherapeutica. 1987;5(2):69-75. PMID 2889217
- [Result] Product Information: Polaramine(R), dexchlorpheniramine maleate. Schering Corporation, Kenilworth, NJ, 1990.
- [Result] Simons FE, Simons KJ, Chung M, Yeh J. The comparative pharmacokinetics of H1-receptor antagonists. Ann Allergy. 1987 Dec;59(6 Pt 2):20-4. PMID 2892445
- [Result] Micromedex novembro de 2015: fenilefrina
- [Result] Hatton RC, Winterstein AG, McKelvey RP, Shuster J, Hendeles L. Efficacy and safety of oral phenylephrine: systematic review and meta-analysis. Ann Pharmacother. 2007 Mar;41(3):381-90. doi: 10.1345/aph.1H679. Epub 2007 Jan 30. PMID 17264159
- [Result] Hengstmann JH, Goronzy J. Pharmacokinetics of 3H-phenylephrine in man. Eur J Clin Pharmacol. 1982;21(4):335-41. doi: 10.1007/BF00637623. PMID 7056280
- [Result] Product Information: phenylephrine hydrochloride injection solution, phenylephrine hydrochloride injection solution. PARENTA Pharmaceuticals, Inc, West Columbia, SC.
- [Result] Micromedex novembro de 2015: cafeína
- [Result] Abbott PJ. Caffeine: a toxicological overview. Med J Aust. 1986 Nov 17;145(10):518-21. doi: 10.5694/j.1326-5377.1986.tb139455.x. PMID 3534532
- [Result] Bula Resfenol - Laboratorios Kleyhertz (Data da bula: 21/05/2014).
- [Result] Brochura Coristina d - Hypermarcas AS.
- [Result] Bertolazi NA. Tradução, adaptação cultural e validação de dois instrumentos de avalição do sono: escala de sonolência de Epworth e Índice de Qualidade de Sono de Pittsburgh. Tese de Mestrado apresentada a UFRGS em 2008. Porto Alegre - RS.
- [Result] Chow, Shao and Wang. Sample Size Calculations. In Clinical Research. Taylor & Francis, NY. (2003): Página 88.
- [Result] Salisbury-Afshar E. Oral antihistamine/decongestant/analgesic combinations for the common cold. Am Fam Physician. 2012 Nov 1;86(9):812-3. No abstract available. PMID 23113460
- [Result] Pinto VF. Estudos clínicos de não-inferioridade: fundamentos e controvérsias. J Vasc Bras; 2010, v.9, n.3.